CLINICAL TRIAL: NCT06299085
Title: Clinical-functional Effects of Bariatric Surgery on the Musculoskeletal System in Relation to the Modification of Body Composition and Bone Turnover After Surgery.
Brief Title: Clinical-functional Effects of Bariatric Surgery on the Musculoskeletal System in Relation to Bone Turnover.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OSTEO-BS (L4191)
Record Dates: First submitted 2024-02-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-11

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: The minimum sample size was determined by considering the circulating levels of gastro-entero hormones (PYY, ghrelin, GLP-1, GIP), adipokines (leptin and adiponectin) and hormones associated with the anabolism of muscle and bone tissue (insulin). as primary endpoints; the highest calculated sample size obtained for ghrelin levels was used for the purposes of this study.
  The calculation was performed using G*Power software (v3.1.9.7) assuming a type I error (α error) of 0.05, a Power (1-β error) of 0.8, an effect size of 0.44.
  The resulting minimum sample size is 42 patients. Taking into account the presence of any drop-outs, 20% more patients will be considered, for a total of 50 patients to be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 50 adult patients suffering from severe or morbid obesity (Other): 50 adult patients suffering from severe or morbid obesity (BMI ≥ 35 kg/m2 in the presence of comorbidities and BMI ≥ 40 kg/m2, respectively), male and female, candidates for bariatric surgery (Sleeve Gastrectomy and Roux-en-Y Gastric Bypass).
  Two timepoints: T0 (pre-hospitalization) and T1 (follow-up 12 months +/- 1 month).
  Expected assessments at T0 and T1:
  * Blood chemistry tests to monitor metabolic markers involved in dietary and metabolic changes.
  * Bone densitometry for body composition analysis (DEXA).
  * Analysis of pre-intervention walking and the ability to recover motor activity after bariatric surgery using gait analysis.
  Interventions: Other: 50 adult patients suffering from severe or morbid obesity, male and female, candidates for bariatric surgery.

INTERVENTIONS:
Other: 50 adult patients suffering from severe or morbid obesity, male and female, candidates for bariatric surgery. — 50 adult patients suffering from severe or morbid obesity (BMI ≥ 35 kg/m2 in the presence of comorbidities and BMI ≥ 40 kg/m2, respectively), male and female, candidates for bariatric surgery (Sleeve Gastrectomy and Roux-en-Y Gastric Bypass).
  Two timepoints: T0 (pre-hospitalization) and T1 (follow-up 12 months +/- 1 month).
  Expected assessments at T0 and T1:
  * Blood chemistry tests to monitor metabolic markers involved in dietary and metabolic changes.
  * Bone densitometry for body composition analysis (DEXA).
  * Analysis of pre-intervention walking and the ability to recover motor activity after bariatric surgery using gait analysis.

SUMMARY:
By studying "in vivo" new possible predictive factors of increased bone turnover and risk of fractures after bariatric surgery, our study aims to improve health not only musculoskeletal but general of patients with severe obesity, a pathology which represents one of the main causes of disability and mortality.

DETAILED DESCRIPTION:
To date, there are no studies in scientific literature aimed at identifying the hormonal mechanisms that could contribute to increased bone turnover in patients undergoing bariatric surgery. All randomized controlled trials conducted to date have focused on nutritional factor deficiency (vitamin D3, calcium and protein), mechanical unloading and reduction of adiposity at the bone marrow level.

By studying "in vivo" new possible predictive factors of increased bone turnover and risk of fractures after bariatric surgery, our study aims to improve health not only musculoskeletal but general of patients with severe obesity, a pathology which represents one of the main causes of disability and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 60 years.
* BMI (Body Mass Index: expressed as weight ratio in kg/height in m2) ≥ 35 kg/m2 with comorbidities or BMI ≥ 40 Kg/m2 without comorbidities.
* Absence of diagnosis of primary obesity.
* Absence of medical-psychiatric contraindications.
* Previous diet therapy and/or pharmacological history verified.
* Signing of the informed consent for the study.
* Patients who are clinical candidates for bariatric surgery (Sleeve Gastrectomy and Roux-en-Y Gastric Bypass).

Exclusion Criteria:

* Presence of chronic diseases of the digestive system, such as chronic intestinal diseases, malabsorption syndrome, diverticulosis of the colon.
* Current pregnancy and/or breastfeeding via self-declaration.
* Subjects suffering from endocrine pathologies (e.g. Cushing's disease, uncontrolled thyroid disease).
* Presence of known renal insufficiency or creatinine levels above 1.8 mg/dl and eGFR < 60 ml/min.
* Presence of chronic liver disease or ALT and AST levels above two standard deviations from normal levels.
* Presence of malignant pathology.
* Alcohol or drug abuse.
* Previous bariatric surgery.
* Severe psychological-psychiatric disorders.
* Difficulty adhering to the protocol due to language barriers or other reasons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Study of new predictive markers of possible bone remodeling through specific blood tests before (pre-admission) and 12 months after bariatric surgery. | Two timepoints: pre-admission before bariatric surgery and 12 months after.
  Study of new predictive markers of possible bone remodeling through specific blood tests before (pre-admission) and 12 months after bariatric surgery by evaluating the circulating levels of gastro-entero hormones, adipokines and hormones associated with anabolism of muscle and bone tissue.

SECONDARY OUTCOMES:
Evaluation of the bone health status of patients pre- and post-bariatric surgery using different methods. | Two timepoints: pre-admission before bariatric surgery and 12 months after.
  Analysis of circulating levels of hormones linked to the anabolism of muscle and bone tissue such as estrogens, androgens and insulin.
  Evaluation of the bone health status of patients pre- and post-bariatric surgery through:
  1. Dual-Energy x-Ray (DEXA) for body composition analysis;
  2. measurement of biomarkers of bone turnover and parathyroid hormone levels;
  3. evaluation of the nutritional status of patients.
  Analysis of pre-intervention walking and the ability to recover motor activity after bariatric surgery using gait analysis. Through Gait Analysis it is possible to analyze body movement and muscle activity.